CLINICAL TRIAL: NCT00240227
Title: The Role of the Alpha 1-adrenergic Antagonist, Prazosin, in the Reduction of Craving and Relapse in Alcohol and Cocaine-dependent Individuals: a Double-blind, Randomized, Controlled Clinical Trial
Brief Title: Prazosin for ETOH or Cocaine Craving
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Experimental procedure did not induce sufficient craving to determine any possible effect of medication.
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REAP 05-0020
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Alcoholism; Cocaine Dependence
Keywords: Alcoholism; Cocaine Dependence; Prazosin; Substance use disorders
MeSH Terms: conditions — Alcoholism; Cocaine-Related Disorders; Substance-Related Disorders | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Other): Placebo no active medication
  Interventions: Drug: placebo
- prazosin (Active Comparator): Prazosin flexible dose titration up to 12 mg per day.
  Interventions: Drug: Prazosin

INTERVENTIONS:
Drug: Prazosin — FDA approved medication for hypertension
  Other Names: Mini Press
  Arms: prazosin
Drug: placebo
  Arms: Placebo

SUMMARY:
This double-blind placebo controlled crossover pilot trial will test the hypothesis that prazosin, an alpha-1 adrenergic receptor antagonist, reduces craving for their drug of choice in cocaine-dependent and alcohol-dependent veterans. Both the study medication period and the placebo period are each 4 weeks in duration.

DETAILED DESCRIPTION:
1. Objective of the project: To evaluate the efficacy of prazosin on the reduction of craving in alcohol and cocaine dependent individuals. The investigators hypothesize that prazosin will be more effective than placebo in the reduction of craving that is stimulated by exposure to visual cues or to intolerance to stress in individuals dependent on cocaine and in individuals dependent on alcohol.

   Specifically, the investigators hypothesize that in this laboratory study:
   * Subjects in the prazosin condition will report a reduction in craving induced in the laboratory by exposure to visual cues compared to subjects in the placebo condition.
   * Subjects in the prazosin condition will show less reaction of the noradrenergic system when craving is induced in the laboratory by exposure to visual cues compared to subjects in the placebo condition.
   * Subjects will be less likely to relapse to their drug of choice while they are in the prazosin condition compared to when they are in the placebo condition. Most individuals who are able to achieve sobriety in chemical dependency treatment eventually relapse. Until the investigators can prevent the cravings for drugs, which usually precedes relapse, it is unlikely that the investigators will have more effective treatment for drug addiction. Our final hypothesis is that the alpha-1, adrenergic antagonist, prazosin, will prove to be an effective pharmacological agent for treatment of drug dependency.
2. Research plan study design: The proposed study will be a double-blind, placebo-controlled, crossover study of prazosin in subjects who are either dependent on alcohol or on cocaine, and who have been able to achieve one month of sobriety while in intensive outpatient treatment. The double-blind, crossover protocol will last 8 weeks and will include 32 subjects; 16 of whom are alcohol-dependent, and 16 of whom are cocaine-dependent. The focus of this first study will be on subjective and physiological measures of craving that will be induced in a controlled setting by exposure to visual cues.
3. Methodology Setting: This study will occur in room 6A-107 in Building 1 at the Veterans Administration Puget Sound Health Care System in Seattle. This is a soundproof room specifically designed and constructed for studies of this type. Participants: 16 alcohol-dependent adults and 16 cocaine-dependent adults presenting for chemical dependency treatment at the VA Puget Sound Health Care System (VAPSHCS) Addiction Treatment Center. Study Procedures: Once potential subjects have provided their consent to participate in the study, they will undergo a 2 hour baseline assessment that consists of some pencil and paper questionnaires, providing a medical and psychiatric history, and a physical exam. They will provide blood for some basic screening labs to insure they are healthy enough to proceed with the study, and have their baseline vital signs measured. Veterans who are screened for the study will then be enrolled once their lab results and the screening process have determined that they do not meet any medical exclusion criteria. At that point, participants will be randomized to either the study medication or placebo. During the course of the study, participants continue with their outpatient chemical dependency treatment through the Addiction Treatment Center at the VA Puget Sound. During the eight weeks of the study, participants will have weekly orthostatic vital sign and adverse events monitoring by the study nurse or physician. All serious or unexpected adverse events will be reported to the FDA and UW Human Subjects Committee in accordance with requirements. Participants will also provide self-reports of drug or alcohol use and urine drug analysis specimens at these weekly visits. At the end of week 4, each participant will be tested in a 1 hour craving session in room 6A-107 at VA Puget Sound. Subjects will have their heart rate and skin conductance response continuously measured, and have their blood pressure measured every 5 minutes. They will be shown 5 1-minute films, 3 of which are designed to be neutral and 2 of which are designed to provoke craving for their drug of choice. They will be asked to complete a subjective scale of craving prior to each video and after the last video. Participants will not be permitted to leave the craving lab after the last film, until they feel that they have subjectively returned to a level of normal physiological arousal and are no longer experiencing any craving.
4. Findings: No findings to date.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Current DSM-IV diagnosis of alcohol dependence or cocaine dependence with no use in last 30 days
* Capacity to provide informed consent
* Actively enrolled in chemical dependency treatment at VA Puget Sound English fluency

Exclusion Criteria:

* Evidence of significant abuse of opiates, PCP, sedatives or anxiolytics
* Suicidal ideation
* DSM IV diagnosis of bipolar mood disorder, schizophrenia or schizoaffective disorder
* Significant acute or chronic medical illness, including unstable angina, recent myocardial infarction, history of congestive heart failure, preexisting hypotension (systolic < 110), or orthostatic hypotension (systolic drop > 20mmHg after two minutes standing or any drop with dizziness), insulin-dependent diabetes mellitus; chronic renal or hepatic failure, pancreatitis, gout, M ni re's disease, benign positional vertigo, narcolepsy
* Concomitant use of alpha-1 antagonists History of prazosin-sensitivity Women who are pregnant, nursing infant(s), or of childbearing potential and not using a contraceptive method judged by the investigator to be effective
* Non-compliance with outpatient chemical dependency treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2004-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. Saxon, MD, Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to one of two sequences, either placebo first or prazosin first. However, the precise numbers of which sequence participants were randomized to are no longer available considering the time (7 years) since the study was completed.
Groups:
- All Study Participants: No active medication
  Prazosin flexible dose titration up to 12 mg per day.
  Prazosin: FDA approved medication for hypertension
Period: Overall Study
Arm/Group | All Study Participants
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Paricipants: No active medication
  Prazosin
  FDA approved medication for hypertension
Arm/Group | All Study Paricipants
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Skin Conductance Response in Response to Provocative Visual Cues Designed to Elicit Craving, Compared to Placebo Group
Time Frame: During lab session
Population: Study was terminated early. No final analyses completed.
Groups:
- Placebo: No active medication
Arm/Group | Placebo | Prazosin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Heart Rate Response in Response to Provocative Visual Cues Designed to Elicit Craving, Compared to Placebo Group
Time Frame: During lab session
Population: Study was terminated early. No final analyses completed.
Arm/Group | Placebo | Prazosin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Blood Pressure Response in Response to Provocative Visual Cues Designed to Elicit Craving, Compared to Placebo Group
Time Frame: During lab session
Population: Study was terminated early. No final analyses completed.
Arm/Group | Placebo | Prazosin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Subjective Experience of Craving in Response to Provocative Visual Cues Designed to Elicit Craving, as Measured by the Within Session Rating for Cocaine/Alcohol Craving
Time Frame: During lab session
Population: Study was terminated early. No final analyses completed.
Arm/Group | Placebo | Prazosin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Self-reports of Substance Use Between Study Medication and Placebo Periods
Time Frame: 4 weeks
Population: Study was terminated early. No final analyses completed.
Arm/Group | Placebo | Prazosin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Urine Drug Analysis Results Between Study Medication and Placebo Periods
Time Frame: 4 weeks
Population: Study was terminated early. No final analyses completed.
Arm/Group | Placebo | Prazosin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Placebo: Placebo no active medication
  placebo
Arm/Group | Placebo | Prazosin
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | Prazosin (N=8)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study procedure intended to induce substance craving failed to induce craving. Thus, any difference between placebo and active medication conditions could not be measured and so the study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes